CLINICAL TRIAL: NCT04202835
Title: A Randomized Pilot Trial Comparing Anti-Thymocyte Globulin (ATG) With ATG Plus Post Transplant Cyclophosphamide (PTCy) for Prophylaxis Against Acute and Chronic Graft Versus Host Disease (GVHD)
Brief Title: ATG Plus PTCy vs ATG for CGVHD Prophylaxis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Cell Therapy Transplant Canada (Unknown); Sanofi (Industry); Ozmosis Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CTTC1901; OZM-099 (Other: Ozmosis Research Inc)
Record Dates: First submitted 2019-11-29; First posted 2019-12-18 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Acute Leukemia; Myelodysplasia; Chronic Graft-versus-host-disease
Keywords: post transplant cyclophosphamide; anti-thymocyte globulin
MeSH Terms: conditions — Anemia, Refractory, with Excess of Blasts; Bronchiolitis Obliterans Syndrome | interventions — Cyclophosphamide; Antilymphocyte Serum; thymoglobulin

STUDY DESIGN:
Intervention Model Description: Randomized pilot trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ATG/PTCy (Experimental): Anti-Thymocyte Globulin (ATG, Thymoglobulin) 4.5 mg/kg IV (divided 0.5, 2.0, 2.0 mg/kg on days -2, -1 and +1); cyclophosphamide (Post Transplant Cyclophosphamide, PTCy) 50 mg/kg IV daily on days +3 and +4.
  Interventions: Drug: Cyclophosphamide; Drug: Anti-Thymocyte globulin (rabbit)
- ATG (Active Comparator): Anti-Thymocyte Globulin (ATG, Thymoglobulin) 4.5 mg/kg IV (divided 0.5, 2.0, 2.0 mg/kg on days -2, -1 and +1).
  Interventions: Drug: Anti-Thymocyte globulin (rabbit)

INTERVENTIONS:
Drug: Cyclophosphamide — Post Transplant Cyclophosphamide
  Arms: ATG/PTCy
Drug: Anti-Thymocyte globulin (rabbit) — Anti-Thymocyte Globulin (rabbit, Thymoglobulin)
  Other Names: Thymoglobulin

SUMMARY:
A Randomized Pilot Trial to test the feasibility of comparing anti-thymocyte globulin plus post transplant cyclophosphamide with anti-thymocyte globulin alone to prevent chronic graft versus host disease.

DETAILED DESCRIPTION:
Patients with acute leukemia or myelodysplastic syndrome will be randomized to receive, or not receive, post transplant cyclophosphamide in addition to anti-thymocyte globulin.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is aged ≥ 16 and deemed medically fit per investigator for protocol
2. The participant has either acute myeloid leukemia in 1st or 2nd complete remission (CR), or has myelodysplastic syndrome
3. The participant will receive a blood progenitor cell graft ("HPC, Apheresis")
4. The participant has a related or unrelated donor, who is fully MHC matched with the recipient at HLA-A, B, C and DRB1.
5. The participant meets the transplant centre's criteria for transplantation, using either myeloablative or reduced intensity conditioning.
6. The participant has good performance status (Karnofsky ≥60%)
7. The participant is able to understand and sign the informed consent form
8. Ability and willingness to comply with study procedures and schedule, in the Investigator's opinion.
9. The participant is receiving their first transplant

Exclusion Criteria:

1. The participant is HIV antibody positive
2. The participant has a hypersensitivity to rabbit proteins or Thymoglobulin® pharmaceutical excipients, glycine or mannitol.
3. The participant has active or chronic infection (i.e. infection requiring oral or IV therapy)
4. The participant (if female and of childbearing potential) is pregnant or breast-feeding at the time of enrollment
5. The participant (if female and of childbearing potential) does not agree to use an adequate contraceptive method from the time of enrollment until a minimum of one year following transplant3
6. The participant (if male and fertile) does not agree to use an adequate contraceptive method from the time of enrollment until a minimum of one year following transplant3
7. The participant has urinary outflow obstruction
8. The participant is in poor condition (determined per institutional guidelines)
9. The participant has acute leukemia in relapse
10. The participant has myelodysplastic syndrome with > 10% marrow blasts
11. The participant is having their second transplant
12. The participant is taking T-cell antibody prophylaxis (anti-CD52)
13. The participant is receiving a cord blood graft or T-cell depleted grafts
14. The participant has mixed phenotype acute leukemia
15. The participant has prior malignancies, except resected nonmelanoma or treated cervical carcinoma in situ. Cancer treated with curative intent ≥ 5 years previously will be allowed. Cancer treated with curative intent < 5 years previously must be reviewed and approved by the sponsors.
16. The participant is in complete remission with incomplete recovery (CRi)

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-10-14 (Actual); Primary Completion 2024-05-18 (Actual); Study Completion 2026-02-07 (Estimated)

PRIMARY OUTCOMES:
Registration of 80 patients within twenty four months | 24 months
  Registration will be documented by the Clinical Research Organization (Ozmosis Research Inc.)

SECONDARY OUTCOMES:
CRFS | 27 months
  Chronic graft versus host disease free- and relapse-free survival (CRFS)
GRFS | 27 months
  Graft versus host disease-, and relapse-, free survival (GRFS)
Survival | 27 months
  Survival (dead/alive) at 100 days for each patient
Complete data collection | 27 months
  The Clinical Research Organization (Ozmosis Research Inc.) will document completeness of data collection
Cost of study | 27 months
  The sponsor (McMaster University) and the Clinical Research Organization (Ozmosis Research Inc.) will compare actual total trial costs in Canadian dollars at trial completion (at completion of outcomes analysis and report) with expected costs as determined for the trial budget.

CONTACTS AND LOCATIONS:
Overall Officials: Irwin R Walker, MBBS, Principal Investigator — McMaster University; Kristjan Paulson, MD, Principal Investigator — CancerCare Manitoba
Locations (9):
- Australia (3):
  - Kinghorn Cancer Centre, St Vincent's Health Network, Darlinghurst, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Australasian Leukaemia and Lymphoma Group, Melbourne, Victoria
- Canada (6):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Juravinski Hospital and Cancer Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Hôpital de l'Enfant-Jésus, Québec, Quebec
  - Saskatchewan Cancer Agency, Saskatoon, Saskatchewan